CLINICAL TRIAL: NCT03658330
Title: Naltrexone Plus Ketamine for the Rapid Treatment of Major Depressive Disorder and Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gihyun Yoon, Principal Investigator, VA Connecticut Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GY0004
Record Dates: First submitted 2018-09-01; First posted 2018-09-05 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Major Depressive Disorder; Alcohol Use Disorder
Keywords: Ketamine; Naltrexone; Depression; Alcohol
MeSH Terms: conditions — Depressive Disorder, Major; Alcoholism; Depression | interventions — Ketamine; Naltrexone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketamine + Naltrexone (Experimental): Subjects will receive (1) intravenous ketamine (0.5 mg/kg) once a week for 4 weeks (a total of 4 infusions) and (2) intramuscular naltrexone (380 mg) once a month (a total of 1 injection).
  Interventions: Drug: Ketamine + Naltrexone

INTERVENTIONS:
Drug: Ketamine + Naltrexone — Subjects will receive (1) intravenous ketamine (0.5 mg/kg) once a week for 4 weeks (a total of 4 infusions) and (2) intramuscular naltrexone (380 mg) once a month (a total of 1 injection).

SUMMARY:
To evaluate if naltrexone plus ketamine is effective in reducing depression and alcohol consumption.

DETAILED DESCRIPTION:
The primary goal of this proposal is to test naltrexone plus repeated ketamine treatment for major depressive disorder and alcohol use disorder in an open-label trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 21-65 years old
2. Current major depressive disorder without psychotic features by DSM-5
3. Montgomery-Åsberg Depression Rating Scale (MADRS) ≥ 20
4. Current alcohol use disorder by DSM-5
5. Heavy drinking at least 3 times in the past month ('heavy drinking' defined as ≥ 5 standard drinks per day for men and ≥ 4 standard drinks per day for women)
6. Abstinence from alcohol drinking for > 5 days prior to ketamine infusion
7. Able to provide written informed consent

Exclusion Criteria:

1. Current substance use disorder by DSM-5 in the past 3 months (except alcohol, tobacco, or cannabis)
2. Current or past history of psychotic features or psychotic disorder
3. Current or past history of delirium or dementia
4. Current uncontrolled hypertension (systolic BP > 170 mm Hg or diastolic BP > 100 mm Hg)
5. Unstable medical condition or allergy to ketamine, naltrexone, or lorazepam---clinically determined by a physician
6. Imminent suicidal or homicidal risk
7. Pregnant or nursing women, positive pregnancy test, or inadequate birth control methods in women of childbearing potential
8. Positive opioid or illicit drug screen test (except marijuana)
9. Opioid use within 10 days prior to study medication (injectable naltrexone) or risks for opioid use during the study
10. Liver enzymes that are three times higher than the upper limit of normal

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Response in symptoms of depression as measured by the Montgomery-Asberg Depression Rating Scale (MADRS) | Day 21
  Response is defined as a ≥ 50% improvement from baseline in MADRS scores. The MADRS has a total range of 0-60. Higher scores represent a worse outcome (i.e., more depression).

SECONDARY OUTCOMES:
Obsessive Compulsive Drinking Scale (OCDS) | Day 21
  The Obsessive Compulsive Drinking Scale is designed to assess alcohol craving and consumption. The scale has a total score range of 0-56. Higher scores represent a worse outcome (i.e., more alcohol problems).

CONTACTS AND LOCATIONS:
Overall Officials: Gihyun Yoon, MD, Principal Investigator — VA Connecticut Healthcare System